CLINICAL TRIAL: NCT05817656
Title: Precise Administration of Sucralfate Powder in Prevention of Delayed Polypectomy Bleeding: a Randomized Clinical Trial
Brief Title: Colonoscopic Sucralfate Spray in Prevention of Delayed Polypectomy Bleeding
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-BR-111-085
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-04

CONDITIONS: Bleeding
Keywords: Polypectomy bleeding; Sulcralfate; Colonoscopic spray
MeSH Terms: conditions — Hemorrhage | interventions — Sucralfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): After polypectomy with a suitable method, either cold snare polypectomy, hot snare polypectomy, endoscopic mucosal resection, or endoscopic submucosal dissection, we will monitor if immediate polypectomy bleeding occurs. If immediate bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine, heater probe coagulation, and/or hemoclipping. If there is no immediate bleeding, we will apply prophylactic clipping in high-risk patients with polyp size ≥ 1cm. After then, we will spray 3g of sucralfate powder through colonoscopy precisely on the polypectomy wound in the intervention group.
  Interventions: Drug: Sucralfate
- Control group (No Intervention): After polypectomy with a suitable method, either cold snare polypectomy, hot snare polypectomy, endoscopic mucosal resection, or endoscopic submucosal dissection, we will monitor if immediate polypectomy bleeding occurs. If immediate bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine, heater probe coagulation, and/or hemoclipping. If there is no immediate bleeding, we will apply prophylactic clipping in high-risk patients with polyp size ≥ 1cm.

INTERVENTIONS:
Drug: Sucralfate — 3g of sucralfate powder through colonoscopy will be sprayed precisely on the polypectomy wound in the intervention group
  Arms: Intervention group

SUMMARY:
Background： Colonoscopy can detect colon polyps and perform excision to the polyps to prevent colon cancer. However, polypectomy bleeding is one of the complications to be noticed, which has an occurrence rate of about 0.4%. Polypectomy bleeding is divided into two types, immediate and delayed bleeding. While immediate polypectomy bleeding can be treated with endoscopic hemostasis during the exam session, delayed polypectomy bleeding occurs a few hours or days after the colonoscopy exam. Patients who encountered delayed polypectomy bleeding usually presented to the hospital for hematochezia, symptoms of anemia, and even hemodynamic instability and end-organ damage. Cold snare polypectomy and prophylactic clipping can reduce the bleeding risk. However, delayed polypectomy bleeding still occurs in high-risk patients, e.g., larger polyps ≥ 1cm. Sucralfate is used for peptic ulcer treatment. It can become a protective layer on the wound to prevent environmental injury. Sucralfate can be used to treat colon ulcers, colitis, and radiation colitis. Whether sucralfate can prevent polypectomy wounds from delayed bleeding is unknown.

Aim： This study aimed to investigate whether precise sucralfate administration on polypectomy wounds can prevent the wound from delayed bleeding.

Method： This is a randomized clinical trial. The study will recruit 160 patients. After randomization, 80 patients will be classified into the intervention group and 80 into the control group. The participants will receive an endoscopic survey as routine, and we will enroll all patients with polyp size ≥ 0.5 cm after polyp excision. Exclusion criteria include patients with an allergy to sucralfate. If immediate polypectomy bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine, heater probe coagulation, and/or hemoclipping. If there is no immediate bleeding, we will apply prophylactic clipping in high-risk patients with polyp size ≥ 1cm. After then, we will spray 3g of sucralfate powder through colonoscopy precisely on the polypectomy wound in the intervention group. All enrolled patients will be monitored for delayed bleeding for 28 days after the colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is the gold standard for the detection of colon polyps for cancer prevention. Colonoscopic polypectomy with the snare is an effective and safe procedure. However, polypectomy bleeding has about a 0.4 % event rate. Polypectomy bleeding can be divided into two types- immediate or delayed polypectomy bleeding. Immediate polypectomy bleeding occurs right after the polyp excision, which can be detected right away with endoscopic hemostasis treatment. Old age ≥ 65 years, comorbid cardiovascular or chronic kidney disease, antiplatelet or anticoagulant agents use, polyp size > 1 cm, laterally spreading polyp, and thick polyp stalk was related to an increased risk of immediate polypectomy bleeding. In contrast, delayed polypectomy bleeding occurs hours or days after the polypectomy. Polyp size > 1 cm, antiplatelet or anticoagulant agents use, the occurrence of immediate polypectomy bleeding, and polyps at the right colon are known risk factors for delayed polypectomy bleeding. An increased size of polyp for every 1 mm significantly increased bleeding by 13%5. Patients who encountered delayed polypectomy bleeding usually presented to the hospital for hematochezia, symptoms of anemia, and even hemodynamic instability and end-organ damage. A polypectomy bleeding-related mortality related was reported at about 0.08%.

At National Cheng Kung University Hospital, we analyzed about 20000 patients underwent colon polypectomy from 2010/01/01 to 2022/07/31. A total of 71 patients encountered delayed polypectomy bleeding, and 29 patients (41%) were with colon polyp size between 0.5 - 1 cm. Polyps with size ≥ 0.5 cm were all at risk of delayed polypectomy bleeding. How to prevent delayed polypectomy bleeding is an important issue for both endoscopists and patients.

Regarding the method of polypectomy, a systemic review and meta-analysis pointed out that cold snare polypectomy was with a lower delayed bleeding risk than hot snare polypectomy. However, only colon polyps ≤ 1 cm were preferred candidates for cold snare polypectomy. Wound closure with clipping after polypectomy is another method to reduce the risk of delayed polypectomy bleeding. For colon polyps > 2 cm in diameter, prophylactic clipping after polypectomy reduces the incidence rate of delayed bleeding. For colon polyps < 2 cm in diameter, prophylactic clipping was not associated with delayed bleeding occurrence. However, delayed polypectomy bleeding still occurs after clipping.

Sucralfate is a complex of aluminum hydroxide and sucrose octasulfate. Sucralfate dissociates in the acid environment to an anionic form, which can bind to the wound base subsequently. This protective barrier can prevent the wound from further environmental injury. Sucralfate has been widely used for wounds and ulcer treatment, e.g., skin wounds, oral ulcers, peptic ulcers, and colon ulcers. Sucralfate can also improve the clinical response to radiation colitis. With the protective effect of the colon mucosa, sucralfate can cover the polypectomy wound and has the potential to avoid further environmental damage from the colon. However, the effect of sucralfate on the prevention of polypectomy bleeding has not been evaluated. This study aimed to investigate whether the precise sucralfate administration on polypectomy wounds can prevent the wound from delayed bleeding.

ELIGIBILITY:
Inclusion Criteria:

* who accept colonoscopy examinations with polyp size ≥ 0.5 cm for polyp excision

Exclusion Criteria:

* patients with an allergy to sucralfate
* patients rejection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-04-14 (Estimated); Study Completion 2024-04-14 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of delayed polypectomy bleeding | 28 days
  The occurrence of delayed polypectomy bleeding. Delayed polypectomy was classified into standard criteria and extended criteria. Standard criteria of delayed postpolypectomy bleeding was defined as emergency attendance, hospitalisation, or need for re-intervention. Extended criteria was defined as blood in stool two days after procedure with or without spontaneous remission.

SECONDARY OUTCOMES:
Incidence rate of need of TAE or surgery | 28 days
  polypectomy wound bleeding requiring transarterial embolization or emergency surgery
length of hospitalization | 28 days
  length of hospitalization due to polyepctomy bleeding
all-cause mortality | 28 days
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Zhang Lin, M.D., Study Director — National Cheng Kung University
Locations (1):
- Hsueh-Chien Chiang, Tainan, Other (Non U.s.), Taiwan

IPD SHARING:
Plan to Share IPD: Yes
After study completed and paper published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years

REFERENCES:
- [Result] Wang YW, Chen HH, Wu MS, Chiu HM; Taiwanese Nationwide Colorectal Cancer Screening Program. Current status and future challenge of population-based organized colorectal cancer screening: Lesson from the first decade of Taiwanese program. J Formos Med Assoc. 2018 May;117(5):358-364. doi: 10.1016/j.jfma.2017.09.010. Epub 2017 Oct 5. PMID 28988890
- [Result] Derbyshire E, Hungin P, Nickerson C, Rutter MD. Post-polypectomy bleeding in the English National Health Service Bowel Cancer Screening Programme. Endoscopy. 2017 Sep;49(9):899-908. doi: 10.1055/s-0043-113442. Epub 2017 Jul 28. PMID 28753697
- [Result] Kim HS, Kim TI, Kim WH, Kim YH, Kim HJ, Yang SK, Myung SJ, Byeon JS, Lee MS, Chung IK, Jung SA, Jeen YT, Choi JH, Choi KY, Choi H, Han DS, Song JS. Risk factors for immediate postpolypectomy bleeding of the colon: a multicenter study. Am J Gastroenterol. 2006 Jun;101(6):1333-41. doi: 10.1111/j.1572-0241.2006.00638.x. PMID 16771958
- [Result] Zhang Q, An Sl, Chen Zy, Fu FH, Jiang B, Zhi Fc, Bai Y, Gong W. Assessment of risk factors for delayed colonic post-polypectomy hemorrhage: a study of 15553 polypectomies from 2005 to 2013. PLoS One. 2014 Oct 1;9(10):e108290. doi: 10.1371/journal.pone.0108290. eCollection 2014. PMID 25271734
- [Result] Buddingh KT, Herngreen T, Haringsma J, van der Zwet WC, Vleggaar FP, Breumelhof R, Ter Borg F. Location in the right hemi-colon is an independent risk factor for delayed post-polypectomy hemorrhage: a multi-center case-control study. Am J Gastroenterol. 2011 Jun;106(6):1119-24. doi: 10.1038/ajg.2010.507. Epub 2011 Jan 25. PMID 21266961
- [Result] Park SK, Seo JY, Lee MG, Yang HJ, Jung YS, Choi KY, Kim H, Kim HO, Jung KU, Chun HK, Park DI. Prospective analysis of delayed colorectal post-polypectomy bleeding. Surg Endosc. 2018 Jul;32(7):3282-3289. doi: 10.1007/s00464-018-6048-9. Epub 2018 Jan 17. PMID 29344790
- [Result] Hassan C, Repici A, Sharma P, Correale L, Zullo A, Bretthauer M, Senore C, Spada C, Bellisario C, Bhandari P, Rex DK. Efficacy and safety of endoscopic resection of large colorectal polyps: a systematic review and meta-analysis. Gut. 2016 May;65(5):806-20. doi: 10.1136/gutjnl-2014-308481. Epub 2015 Feb 13. PMID 25681402
- [Result] Shinozaki S, Kobayashi Y, Hayashi Y, Sakamoto H, Lefor AK, Yamamoto H. Efficacy and safety of cold versus hot snare polypectomy for resecting small colorectal polyps: Systematic review and meta-analysis. Dig Endosc. 2018 Sep;30(5):592-599. doi: 10.1111/den.13173. Epub 2018 May 14. PMID 29675857
- [Result] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Result] Qu J, Jian H, Li L, Zhang Y, Feng B, Li Z, Zuo X. Effectiveness and safety of cold versus hot snare polypectomy: A meta-analysis. J Gastroenterol Hepatol. 2019 Jan;34(1):49-58. doi: 10.1111/jgh.14464. Epub 2018 Sep 26. PMID 30176072
- [Result] Matsumoto M, Kato M, Oba K, Abiko S, Tsuda M, Miyamoto S, Mizushima T, Ono M, Omori S, Takahashi M, Ono S, Mabe K, Nakagawa M, Nakagawa S, Kudo T, Shimizu Y, Sakamoto N. Multicenter randomized controlled study to assess the effect of prophylactic clipping on post-polypectomy delayed bleeding. Dig Endosc. 2016 Jul;28(5):570-6. doi: 10.1111/den.12661. Epub 2016 May 25. PMID 27018874
- [Result] Boumitri C, Mir FA, Ashraf I, Matteson-Kome ML, Nguyen DL, Puli SR, Bechtold ML. Prophylactic clipping and post-polypectomy bleeding: a meta-analysis and systematic review. Ann Gastroenterol. 2016 Oct-Dec;29(4):502-508. doi: 10.20524/aog.2016.0075. Epub 2016 Jul 28. PMID 27708518
- [Result] Turan AS, Pohl H, Matsumoto M, Lee BS, Aizawa M, Desideri F, Albeniz E, Raju GS, Luba D, Barret M, Gurudu SR, Ramirez FC, Lin WR, Atsma F, Siersema PD, van Geenen EJM; Prophylactic Clipping Collaborative Group. The Role of Clips in Preventing Delayed Bleeding After Colorectal Polyp Resection: An Individual Patient Data Meta-Analysis. Clin Gastroenterol Hepatol. 2022 Feb;20(2):362-371.e23. doi: 10.1016/j.cgh.2021.05.012. Epub 2021 May 12. PMID 33991691
- [Result] Nagashima R. Mechanisms of action of sucralfate. J Clin Gastroenterol. 1981;3(Suppl 2):117-27. PMID 6798100
- [Result] Masuelli L, Tumino G, Turriziani M, Modesti A, Bei R. Topical use of sucralfate in epithelial wound healing: clinical evidences and molecular mechanisms of action. Recent Pat Inflamm Allergy Drug Discov. 2010 Jan;4(1):25-36. doi: 10.2174/187221310789895649. PMID 19832693
- [Result] Ala S, Saeedi M, Janbabai G, Ganji R, Azhdari E, Shiva A. Efficacy of Sucralfate Mouth Wash in Prevention of 5-fluorouracil Induced Oral Mucositis: A Prospective, Randomized, Double-Blind, Controlled Trial. Nutr Cancer. 2016;68(3):456-63. doi: 10.1080/01635581.2016.1153666. Epub 2016 Mar 23. PMID 27007594
- [Result] Hunt RH. Treatment of peptic ulcer disease with sucralfate: a review. Am J Med. 1991 Aug 8;91(2A):102S-106S. doi: 10.1016/0002-9343(91)90459-b. PMID 1882894
- [Result] Fernandez OOA, Pereira JA, Campos FG, Araya CM, Marinho GE, Novo RS, Oliveira TS, Franceschi YT, Martinez CAR. EVALUATION OF ENEMAS CONTAINING SUCRALFATE IN TISSUE CONTENT OF MUC-2 PROTEIN IN EXPERIMENTAL MODEL OF DIVERSION COLITIS. Arq Bras Cir Dig. 2017 Apr-Jun;30(2):132-138. doi: 10.1590/0102-6720201700020012. PMID 29257850
- [Result] McElvanna K, Wilson A, Irwin T. Sucralfate paste enema: a new method of topical treatment for haemorrhagic radiation proctitis. Colorectal Dis. 2014 Apr;16(4):281-4. doi: 10.1111/codi.12507. PMID 24299100
- [Result] Kochhar R, Sriram PV, Sharma SC, Goel RC, Patel F. Natural history of late radiation proctosigmoiditis treated with topical sucralfate suspension. Dig Dis Sci. 1999 May;44(5):973-8. doi: 10.1023/a:1026612731210. PMID 10235606
- [Derived] Chiang HC, Chen PJ, Yang EH, Kuo TL, Hsieh MT, Kang JW, Cheng HC, Chang WL, Chen WY, Chiu HC, Lin MY, Hong TC, Chiang CM, Chen WC, Huang KK, Lu MH, Wu MH, Chen CY, Lin XZ, Chuang CH. Clinical Trial: Precise Administration of Sucralfate Powder in Prevention of Delayed Postpolypectomy Bleeding. A Randomized Controlled Trial. Clin Transl Gastroenterol. 2025 Apr 1;16(4):e00818. doi: 10.14309/ctg.0000000000000818. PMID 39836033